CLINICAL TRIAL: NCT04845282
Title: Effects of Graded Protein Intake and Resistance Training on Body Composition in Older Adults
Brief Title: Effects of Graded Protein Intake on Body Composition in Older Adults
Acronym: GPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Gary Miller, Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00024112
Record Dates: First submitted 2021-04-05; First posted 2021-04-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenia
Keywords: Protein; Skeletal Muscle; Body Composition; Ultrasonography; Resistance Training
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups. The first group will consume a set schedule of additional dietary protein, while the second group will consume a diet with the recommended dietary allowance of protein.
Who Masked: Investigator
Masking Description: Participants will be aware of their intervention, but the primary investigator and research staff performing assessments will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Graded Protein plus Resistance Training (Experimental): This group will participate in a progressive resistance training program and will be instructed to consume a diet with a gradation of protein over the 12 week study duration.
  Interventions: Dietary Supplement: Graded Protein plus Resistance Training
- RDA Protein plus Resistance Training (Active Comparator): This group will participate in a progressive resistance training program and will be instructed to consume a diet with the recommended daily allowance of protein over the 12 week study duration.
  Interventions: Dietary Supplement: RDA Protein plus Resistance Training

INTERVENTIONS:
Dietary Supplement: Graded Protein plus Resistance Training — Participants will be counseled to consume the specific level of dietary protein plus the protein supplement is MusclePharm Combat 100% Whey. Specific values per week are listed below:
  Week 1: 25 g of protein supplement (0.8 g protein/kg body weight) Week 2: 25 g of protein supplement (1.0 g protein/kg body weight) Week 3: 50 g of protein supplement (1.2 g protein/kg body weight) Week 4: 50 g of protein supplement (1.4 g protein/kg body weight) Week 5: 50 g of protein supplement (1.4 g protein/kg body weight) Week 6: 75 g of protein supplement (1.6 g protein/kg body weight) Week 7: 75 g of protein supplement (1.8 g protein/kg body weight) Week 8: 75 g of protein supplement (2.0 g protein/kg body weight) Week 9: 75 g of protein supplement (2.2 g protein/kg body weight) Week 10: 100 g of protein supplement (2.2 g protein/kg body weight)
  Arms: Graded Protein plus Resistance Training
Dietary Supplement: RDA Protein plus Resistance Training — Participants will be counseled to consume the RDA level of protein (0.8g/kg/day) utilizing only dietary protein.
  Arms: RDA Protein plus Resistance Training

SUMMARY:
This clinical trial is intended to evaluate the effects of protein intake graded to resistance training volume over a 10-week period on macroscopic skeletal muscle adaptations and body composition. Briefly, all participants will complete a progressive resistance training protocol for 10 weeks, with one group consuming a constant amount of total daily protein (RDA of 0.8g/kg/day) to serve as an active comparator. The alternative group will consume total daily protein and protein supplement in a graded manner designed to increase as overall training volume increases. Protein intake and resistance training protocols are described in full elsewhere. The investigators hypothesize that the graded protein intake group will see larger benefits to skeletal muscle function, size, and body composition than the active comparator.

DETAILED DESCRIPTION:
It is well established that aging induces a loss of skeletal muscle across a lifespan. The two primary considerations in attenuating this loss of skeletal muscle are nutritional intake, specifically protein consumption, and physical activity levels, specifically resistance training. Both of these factors have been shown to improve skeletal muscle adaptation outcomes in older adults. One primary consideration in the skeletal muscle loss in older adults is the concept of anabolic resistance, suggesting that older adults require a greater amount of protein consumption to elicit similar rates of muscle protein synthesis as compared to their younger counterparts. From this study, the investigators hope to reveal the effect between protein intake graded to resistance training vs constant protein intake at the recommended daily allowance in conjunction with the same resistance training protocol on body composition. The purpose of this study is to examine the skeletal muscle adaptations that occur in older adults consuming protein graded to resistance training volume as compared to older adults who consume protein at a constant level while resistance training (RT). Our hypotheses are:

1. Protein intake graded to RT volume will enhance skeletal muscle adaptation in older adults to a greater degree than those consuming protein at a constant rate, as measured via lean soft tissue mass assessed by dual energy x-ray absorptiometry (DXA)
2. Older adults consuming protein graded to RT volume will enhance strength to a greater degree than those consuming protein at a constant rate, as measured via isokinetic dynamometry and 3 repetition maximums of select exercises.
3. Older adults consuming protein graded to RT volume will see a greater change in muscle tissue thickness compared to those consuming protein at a constant rate, as measured via muscular ultrasound.

Community dwelling older adults (>55 years; men and women) who have not adhered to a progressive RT program in the last 3 months will be recruited for participation in this pilot study (n=20). All women recruited will be post-menopausal. In an initial telephone screening, participants will be assessed for eligibility criteria, and it will also be determined whether they are willing to be randomized into either of the two groups. The requirements of each intervention group will be explained in detail. Participants will be assessed for willingness to make necessary alterations to their diet, willingness to adhere to RT protocol, and willingness to consume the necessary amount of protein supplement. Once participants are recruited, they will be subsequently randomized using a web based program (https://www.randomlists.com/team-generator) wherein group assignments will be placed in numbered envelopes and opened by an independent researcher. This will be used to randomize participants to one of the two experimental groups. This randomization and assignment will be completely random, and not stratified to any subset of variables. All groups will complete the same resistance training protocol. Overall study design, resistance training protocol, detailed nutritional protocols are outlined in the tables submitted in supporting documents. Briefly, all participants will be assigned a 10-week RT protocol, adhering to the 2009 Position Stand from the American College of Sports Medicine, based on their baseline tested 3 repetition maximums. Participants in the graded protein intake group will be provided a certain amount of Whey Protein (WP) supplement to consume post-training session on training days, and between meals on non-training days. The control group will not receive WP supplement, whereas the intervention group will receive 25 g of WP supplement per day beginning at week 1 and will progress to 75g of WP supplement/day by week 10 of the intervention. This supplementation will assist overall protein intake, as the control group will consume a constant 0.8g/kg/day throughout the course of the study and the intervention group will consume 0.8 g/kg/day at week 1 and progress to 2.2 g/kg/day at week 10. For example, an 80 kg individual will consume a total of 176 g of protein/day at week 10, with 75 g of this protein coming from supplementation, and the additional 76g coming from dietary intake throughout the day. Should prescribed supplementation exceed the 2.2 g/kg/day threshold, adjustments will be made in protocol to accommodate proper protein intake. The investigators expect no adverse effects on renal and liver function as a result of increased protein intake based on the findings of a recent meta analysis by Devries et al. (2018). Additionally, participants will consume a ~500 kcal surplus per day to ensure adequate energy for protein accretion and recovery.

Covid-19 Protocol:

Investigators, study staff, and participants alike share responsibility for the health and safety of each other in an exercise/testing space. Maintaining a consistent six feet of distance; wearing face coverings that cover our mouths and noses; limiting our gathering sizes; and isolating or quarantining when ill or exposed to someone with the virus are Wake Forest University directives and policies investigators, study staff, and participants all must follow. Participants are encouraged to visit Our Way Forward to stay informed about the latest guidance and stay up to date regarding public health policy. The study team will follow guidelines set forth by public health officials.

Specifically, in this study, investigators, staff, and participants will mitigate the risks of virus transfer and take care of our community by abiding by the following safety directives:

* maintain six feet of distance at all times when feasible.
* wear a face covering for the entirety of time indoors and out. This face covering should cover your mouth and your nose, and adhere to our University face covering policy (no face shields without masks; no neck gaiters; no bandanas; and no masks, including N95, with a one-way valve).
* stay out of sessions when sick or after being exposed to someone who is sick.

In this study, any participant who does not follow these requirements will be asked to follow the safety directives.

Participants will be offered a mask should they not have one.

If participants do not comply, they will be asked to leave the study space out of an abundance of caution in regard to other participants and study staff.

ELIGIBILITY:
Inclusion Criteria:

* >55 years of age
* Able to provide transportation to resistance training sessions and data collection days
* Able to read and write in English
* Have not adhered to a progressive resistance training program in the past three months
* Able to ambulate without assistance
* Willingness to provide informed consent and participate in the intervention
* Do not have a comorbidity that could be exacerbated by study protocol, such as severe cardiovascular disease, type I or type II diabetes, renal failure, liver disorders, or thyroid disease OR can provide explicit written consent from a primary care physician indicating that they can participate in this study.

Exclusion Criteria:

* Currently consuming an agent known to be confounding to skeletal muscle adaptation, such supplements that include, but are not limited to creatine monohydrate, growth hormone, or testosterone replacement therapy
* Currently undergoing cancer treatment
* Used whey protein supplements within the past three months
* Pre-menopausal status for women

Ages: 55 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Whole body lean soft tissue mass (kg) from baseline to 10 weeks | Baseline and 10 weeks
  Lean soft tissue mass (LSTM) will be assessed via dual-energy X-ray absorptiometry (DXA) (GE Lunar iDXA) both pre- and post-intervention. Scans will be performed at the same time of day (0600-1300), in a fasted state (>10 hrs fasted), and at least 72 hours after the final bout of training to account for cellular edema at baseline and after 10 wk of intervention on participants wearing general sports attire. Participants will remain supine and aligned with the scanner table as prescribed by the manufacturer. Data from DXA scans will include total body lean soft tissue mass in kilograms as assessed by the accompanying software. Testing will occur at the Wake Forest University Worrell Professional Center (HES) in the Body Composition Laboratory.
Change in Whole body fat mass (kg) from baseline to 10 weeks | Baseline and 10 weeks
  Lean soft tissue mass (LSTM) will be assessed via dual-energy X-ray absorptiometry (DXA) (GE Lunar iDXA) both pre- and post-intervention. Scans will be performed at the same time of day (0600-1300), in a fasted state (>10 hrs fasted), and at least 72 hours after the final bout of training to account for cellular edema at baseline and after 10 wk of intervention on participants wearing general sports attire. Participants will remain supine and aligned with the scanner table as prescribed by the manufacturer. Data from DXA scans will include total body fat mass in kilograms as assessed by the accompanying software. Testing will occur at the Wake Forest University Worrell Professional Center (HES) in the Body Composition Laboratory.
Change in regional (specifically the lower extremity) lean soft tissue mass (kg) from baseline to 10 weeks | Baseline and week 10
  Lean soft tissue mass (LSTM) will be assessed via dual-energy X-ray absorptiometry (DXA) (GE Lunar iDXA) both pre- and post-intervention. Scans will be performed at the same time of day (0600-1300), in a fasted state (>10 hrs fasted), and at least 72 hours after the final bout of training to account for cellular edema at baseline and after 10 wk of intervention on participants wearing general sports attire. Participants will remain supine and aligned with the scanner table as prescribed by the manufacturer. Data from DXA scans will include lower extremity lean soft tissue mass in kilograms as assessed by the accompanying software. Testing will occur at the Wake Forest University Worrell Professional Center (HES) in the Body Composition Laboratory.
Change in regional (specifically the lower extremity) fat mass (kg) from baseline to 10 weeks | Baseline and week 10
  Lean soft tissue mass (LSTM) will be assessed via dual-energy X-ray absorptiometry (DXA) (GE Lunar iDXA) both pre- and post-intervention. Scans will be performed at the same time of day (0600-1300), in a fasted state (>12 hrs fasted), and at least 72 hours after the final bout of training to account for cellular edema at baseline and after 10 wk of intervention on participants wearing general sports attire. Participants will remain supine and aligned with the scanner table as prescribed by the manufacturer. Data from DXA scans will include lower extremity fat mass in kilograms as assessed by the accompanying software. Testing will occur at the Wake Forest University Worrell Professional Center (HES) in the Body Composition Laboratory.

SECONDARY OUTCOMES:
Change in Muscular Function (3 repetition maximum) from baseline to 5 weeks to 10 weeks | Baseline, Week 5, and Week 10
  3 repetition maximums (RMs) will be assessed at pre-, week 6, and post-intervention as described in Table 1 in the support documentation. 3 RMs will be collected for the bilateral leg press and the bilateral leg extension to be considered for analysis. Participants will complete 3 RM testing under the supervision of trained research staff. Participants will perform three repetitions at a given load and progress at their own pace until endpoints of testing are reached. Endpoints are defined as the inability to complete a given load for 3 repetitions, non-adherence to proper form or full range of motion, or the voluntary cessation of exercise by the participant.
Change in Muscular Function (isokinetic dynamometry) from baseline to 5 weeks to 10 weeks | Baseline, Week 5, Week 10
  Peak Torque will be assessed via isokinetic dynamometry. Participants will be seated and strapped into a Humac NORM isokinetic dynamometer (Computer Sports Medicine Inc., Stoughton, MA) ensuring that their hip angle is ~90 degrees. The input axis of the dynamometer will be aligned with the lateral epicondyle of the left femur. All measures will be taken in the left leg, and will be taken in duplicate. The highest peak torque produced throughout either trial will be used. Dynamometry measures will be taken at pre-, week 6, and post-intervention.
Change in Muscle Tissue Thickness from baseline to 10 weeks | Baseline, Week 10
  Muscle tissue thickness of the vastus lateralis (VL) will be assessed via 6-13 MHz transducer muscular ultrasound (SonoSite M-Turbo), at least 72 hours after completion of the most recent training session. Ultrasonography will take place at the midway point between the iliac crest and the patella of the right femur, with subjects in a supine position. Participants will be instructed to assume a supine position for >10 minutes to account for fluid shifting. Duplicate measures will be taken and the average muscle tissue thickness (MT) will be recorded. Testing will take place at HES in the Pulmonary Function and Ultrasound Laboratory.
Height and weight will be combined to report change in BMI in kg/m^2 from baseline to 5 weeks to 10 weeks | Baseline, Week 5, Week 10
  Height and body mass measures will be collected via wall-mounted stadiometer (Detecto) and digital scale (Tanita) respectively with heights and weights collected to the nearest 0.1 kg and 0.5 cm. Height and weight measures will be used to compute body mass index (BMI) defined as weight in kilograms divided by height in meters squared (kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Miller, Ph.D., Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University Clinical Research Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devries MC, Sithamparapillai A, Brimble KS, Banfield L, Morton RW, Phillips SM. Changes in Kidney Function Do Not Differ between Healthy Adults Consuming Higher- Compared with Lower- or Normal-Protein Diets: A Systematic Review and Meta-Analysis. J Nutr. 2018 Nov 1;148(11):1760-1775. doi: 10.1093/jn/nxy197. PMID 30383278
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- See also: Whey Protein to be used — http://musclepharm.com/products/combat-100-whey-2